CLINICAL TRIAL: NCT04472923
Title: Effect of Biofeedback Training on Functional Non-Retentive Fecal Incontinence in Children
Brief Title: Biofeedback Training Fecal Incontinence in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Mohamed A. Abdel Ghafar, Associate Professor of Physical Therapy, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BatterjeeMC
Record Dates: First submitted 2020-07-07; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Fecal Incontinence in Children
Keywords: Fecal incontinence; Biofeedback; long-term; Children
MeSH Terms: conditions — Fecal Incontinence | interventions — Diet; Exercise; Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: The present study included 100 children of both sexes that were included with an age ranged from (5-14 years) with FNRFI with normal bowel habits, normal defecation frequency, and normal stool consistency with incontinence score ranging from 6-24 according to Vaizey score 12. Exclusion criteria included; children who have traumatic sphincter injury, fecal impaction, spinal diseases causing incontinence, anorectal malformation, and children who were not cooperative. Patients included in this study were randomly divided and allocated into two groups Control group and Study group. Written informed consent was obtained from parents of all included children.
  A detailed history was taken including bowel habits, duration history of trauma. Complete physical examination to exclude patients requiring surgical correction
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients belonging to the control group received conventional physical therapy program in the form of diet and Kegel exercises.
  Interventions: Procedure: Traditional Treatment
- Study group (Experimental): Patients belonging to the study group were subjected to the same conventional physical therapy program in addition to biofeedback training
  Interventions: Device: Biofeedback

INTERVENTIONS:
Procedure: Traditional Treatment — Patients belonging to the control group received conventional physical therapy program in the form of:
  1. Dietetic Regulation: The diet was given in the form of the bulk-forming diet, fruits, vegetables, cereals, and bran.
  2. Pelvic floor muscle exercises (Kegal exercises): The patient was instructed to lie crock lying position with knees bent. He/she was instructed to pull his/her pelvic muscles upward and inward and hold the contraction for 6 seconds as if to hold back a defecation movement, followed by relaxation for 6 seconds. The exercise was repeated 25 times. Gradually increase the time until reaching 10 seconds of contraction and relaxation for each with repetition up to 30 times. The exercises applied twice per week for 3 months.
  Other Names: Diet and exercises
  Arms: Control group
Device: Biofeedback — Patients belonging to the study group were subjected to the same conventional physical therapy program in addition to biofeedback training.
  Biofeedback was planned after full guardians' education. Local hygiene for perianal skin for soiling episodes and using zinc oxide cream to prevent excoriation. Biofeedback was done using two types of catheters; a 24-channel water-perfused catheter with latex balloon for sensory training and a double-lumen rectal PVC balloon clothed catheter (MMS U-72210) for strength training. Each biofeedback session took 30 minutes with two sessions per week for 3 months.
  Arms: Study group

SUMMARY:
Fecal incontinence (FI) is the inability to control bowel movements, causing stool to leak from rectum it ranges from an occasional leakage of stool while passing gas to a complete loss of bowel control after the age of 4 years1. Functional non-retentive fecal incontinence (FNRFI) is fecal incontinence in a child with a mental age of more than 4 years with no evidence of metabolic, inflammatory, or anatomical cause2.

The long-term result of biofeedback therapy is one of the most important subjects of controversy, and few studies have extended to 2 years of follow-up 11. So, the purpose of this study was to evaluate quantitatively the short-term and long-term efficacy of biofeedback training as a treatment tool designed to control functional non-retentive fecal incontinence in children and its long term impact on the quality of life.

DETAILED DESCRIPTION:
Functional non-retentive fecal incontinence (FNRFI) is fecal incontinence in a child with a mental age of more than 4 years with no evidence of metabolic, inflammatory, or anatomical cause2.

It is an extremely embarrassing and psychologically frustrating shameful problem with a bad impact on children3. It can lead to social isolation, loss of self-confidence, depression, and behavioral problems4. The underlying mechanism of functional non-retentive fecal incontinence is largely unknown. The pathophysiology seems to be complex and it is considered to be a multifactorial disorder5. Approximately 95% of the children had no organic cause and these children are considered to have a functional defecation disorder. Of this, in approximately 80% of these children FI is results of constipation and is treated with laxatives, the remaining 20% without signs of fecal retention is classified as FNRFI6 The negative psychological and social impact for these children is high, however, and requires adequate intervention7. Biofeedback therapy is a feasible option that has been used for fecal incontinence over several decades8. The underlying premise of biofeedback, as with learning any physical activity, is that "practice makes perfect" if the learner is provided with accurate feedback to make adjustments to optimize performance So, the purpose of this study was to evaluate quantitatively the short-term and long-term efficacy of biofeedback training as a treatment tool designed to control functional non-retentive fecal incontinence in children and its long term impact on the quality of life.

Methods:

The present study included 100 children of both sexes that were included with an age ranged from (5-14 years) with FNRFI with normal bowel habits, normal defecation frequency, and normal stool consistency with incontinence score ranging from 6-24 according to Vaizey score 12. Exclusion criteria included; children who have traumatic sphincter injury, fecal impaction, spinal diseases causing incontinence, anorectal malformation, and children who were not cooperative. Patients included in this study were randomly divided and allocated into two groups Control group and Study group. Written informed consent was obtained from parents of all included children.

A detailed history was taken including bowel habits, duration history of trauma. Complete physical examination to exclude patients requiring surgical correction.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from (5-14 years) with FNRFI with normal bowel habits
* Children with normal defecation frequency and normal stool consistency
* Children with incontinence score ranging from 6-24 according to Vaizey score

Exclusion Criteria:

* Children who have traumatic sphincter injury.
* Children who have Fecal impaction
* Children who have Spinal diseases causing incontinence
* Children who have Anorectal malformation
* Children who were not cooperative

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-07-05 (Actual)

PRIMARY OUTCOMES:
Number of incontinence episodes | 24 months
  Change in the number of incontinence episodes
Incontinence Score using Vaizey incontinence score | 24 months
  Questionnaire ranging from zero (indicating complete continence) to 24 (indicating total incontinence).

SECONDARY OUTCOMES:
Fecal Incontinence Quality of life Score | 24 months
  Change in quality of life score measured on a scale between 1 and 4, where 1 is very affected and 4 is not affected
Resting pressure (mm hg) | 3 months
  Pressure during relaxation of the anal sphincter
Squeeze pressure (mm hg) | 3 months
  Pressure during contraction of the anal sphincter
First sensation (volume of the balloon by cm water) | 3 months
  First sensation of the stool in the rectum
First Urge (volume of the balloon by cm water) | 3 months
  The patient is trying to hold defecation and he can
Intense urge (volume of the balloon by cm water) | 3 months
  The Patent can no longer control the defecation

CONTACTS AND LOCATIONS:
Overall Officials: Emad M Abdelrahman, M.D., Study Director — Bnha University
Locations (1):
- Benha University, Banhā, Al Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After Publication, the investigators would like to share the data with other researchers who interested in this topic
Supporting Information: Study Protocol
Time Frame: After publication
Access Criteria: Not available now